CLINICAL TRIAL: NCT04500093
Title: Does Capsulectomy, Performed in Total Hip Arthroplasty With a Direct Anterior Approach Cause Knee Extension Strength Loss?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Orkhan Aliyev, MD, Resident Doctor in Orthopaedic Surgery, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24959901
Record Dates: First submitted 2020-08-01; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Coxarthrosis; Muscle Weakness
Keywords: Hip; Arthroplasty; Quadriceps strenght; Muscle Weakness; Knee; Flexion; Extension
MeSH Terms: conditions — Osteoarthritis, Hip; Muscle Weakness | interventions — Wound Healing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsulotomy with Repair (Experimental): Repair after capsulotomy in direct anterior hip arthroplasty
  Interventions: Procedure: Capsulotomy with Repair
- Capsuloectomy (Active Comparator): Capsuloectomy in direct anterior hip arthroplasty
  Interventions: Procedure: Capsuloectomy

INTERVENTIONS:
Procedure: Capsulotomy with Repair — Capsulotomy with Repair
  Arms: Capsulotomy with Repair
Procedure: Capsuloectomy — Capsuloectomy
  Arms: Capsuloectomy

SUMMARY:
Total hip arthroplasty (THA) has been successful in relieving pain and restoring function in patients with advanced arthritis of the hip joint. Increased focus on earlier recovery and decreased postoperative pain has improved overall satisfaction. However, there is still a gap between the clinical scores in objective surveys and patient satisfaction. Direct anterior approach total hip arthroplasty has a low dislocation rate, abductor strength restoration, acceleration, and cosmetic advantages. In this method, capsulotomy with repair or capsulectomy is applied as the preferences of surgeons. Therefore, this can cause both a decrease in hip flexion strength and a loss in knee extension strength. Our aim in this study is to reveal how much muscle loss was caused by comparing both methods with the intact side.

DETAILED DESCRIPTION:
Published data assessing biomechanical performance after THR are sparse. The majority of studies assessing post-THR hip function using robotic dynamometry have focused on evaluating surgical outcomes and prosthetic selection. These studies provide insight regarding the strength deficits of older adults after THR. However, the data are not consistent, making it difficult to assess the nature of the deficit.

ELIGIBILITY:
Inclusion Criteria:

* All primary THA

Exclusion Criteria:

* Secondary THA

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-02 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Muscle Weakness | 1 year
  Newton

SECONDARY OUTCOMES:
Harris Hip Score | 1 year
  Score

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP